CLINICAL TRIAL: NCT05567900
Title: Hungarian Women's Health Care Seeking Behavior and Knowledge of Urinary Incontinence and Pelvic Organ Prolapse
Brief Title: Health Care Seeking Behavior and Knowledge Assessment of Hungarian Women About Pelvic Floor Disorders
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: BMEÜ/379-3/2022/EKU-1
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse; Knowledge, Attitudes, Practice; Behavior, Health
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse; Behavior; Health Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess women's health care seeking behavior and knowledge of urinary incontinence and pelvic organ prolapse and to culturally adapt the Prolapse and Incontinence Knowledge Questionnaire (PIKQ) for the Hungarian population.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age 18 and above
* Ability to read and write Hungarian
* Willing to complete the online survey
* Providing consent to participate

Exclusion Criteria:

* Respondents who had already completed the questionnaire on a prior occasion
* Respondents who unable to complete the online survey due to illiteracy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years or older who are able to read and write Hungarian.
Sampling Method: Non-Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence and pelvic organ prolapse knowledge | Baseline
  The Prolapse and Incontinence Knowledge Questionnaire (PIKQ) is used to assess knowledge. It consists of two distinct scales: the first one measures knowledge about urinary incontinence knowledge, while the second one measures knowledge about pelvic organ prolapse. The total score of each scale can range from 0 to 12. Higher scores indicate greater knowledge.
Health seeking behavior | Baseline
  Participants report whether they have sought health care for urinary incontinence. The outcome is the proportion of participants who have ever sought care, among those who reported a history of urinary incontinence.

SECONDARY OUTCOMES:
Urinary incontinence | Baseline
  The International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF) was used to gather information about the symptoms of urinary incontinence. It contains six questions. The total score can range from 0 to 21. Higher scores indicate more severe symptoms.
Practice of pelvic floor muscle training (PFMT) | Baseline
  The PFMT practice scale of the Pelvic Floor Muscle Training Patient reported Outcome Measures (PFMT-P) was used to assess women's practice of PFMT. Questions dealt with source of knowledge about PFMT, practice and correct performance.

CONTACTS AND LOCATIONS:
Overall Officials: Márta Hock, Habilitation, Study Director — University of Pecs
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No